CLINICAL TRIAL: NCT02078700
Title: Feasibility of an Early Palliative Care Intervention for Metastatic Cancer Patients. A Phase 2 Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CE148/2012
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2015-01

CONDITIONS: Lung Cancer; Mesothelioma; Pancreas Cancer; Gastric Cancer
Keywords: cancer; early palliative care; feasibility
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma; Pancreatic Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- early palliative care programme (Experimental): Patients will be proposed to be followed by the Palliative Care Team
  Interventions: Other: The early palliative care programme

INTERVENTIONS:
Other: The early palliative care programme — The intervention consists of an early integration of a palliative care programme with the standard care performed by the oncologists-pneumologists that are following the cancer patients. The intervention will be delivered by the specialised Palliative Care Unit (PCU) of the hospital. Each patient meets the professionals of the PCU by 30 days by cancer diagnosis and at least monthly thereafter in the outpatint settings.

SUMMARY:
The objective of this phase 2 study is to evaluate the feasibility of an early palliative care intervention for metastatic cancer patients. Feasibility will be assessed in terms of percentage of patients that accept the proposal of the early palliative care intervention and that effectively start to be followed in the palliative care out-patient clinic. The study will be performed in a consecutive series of newly diagnosed patients affected by lung cancer (NSCLC or SCLC, stage IIIb, IV), mesothelioma (stage II, IV), pancreas (stage IV), stomach (stage IIIb-IV).

ELIGIBILITY:
Inclusion Criteria:

* patients within 8 weeks of cancer diagnosis confirmed by histology or cytology
* lung cancer (NSCLC or SCLC) stage IIIb-IV OR mesothelioma stage III-IV OR pancreas cancer stage IV, OR gastric cancer stage IIIb-IV
* age more than 18 years
* performance status (ECOG) ≤ 2;
* ability to read, understand and fill-in the questionnaires
* written informed consent to the study

Exclusion Criteria:

* any chemotherapy, radiotherapy or ormonotherapy for any tumour in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
percentage of cancer patients that accept and attend the early palliative care programme | up to 30 days after the diagnosis of cancer
  percentage of eligible cancer patients that accept the proposal of the intervention (the early palliative care programme) and that, by 30 days after the diagnosis, effectively start to be followed by the Palliative Care Unit

SECONDARY OUTCOMES:
percentage of cancer patients that receive the proposal of early palliative by the oncologists-pneumologists | up to 30 days after the diagnosis of cancer
  percentage of newly diagnosed eligible cancer patients that receive the proposal of the itegrated early palliative care programme

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Arcispedale S.Maria Nuova, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costantini M, Apolone G, Tanzi S, Falco F, Rondini E, Guberti M, Fanello S, Cavuto S, Savoldi L, Piro R, Mecugni D, Di Leo S. Is early integration of palliative care feasible and acceptable for advanced respiratory and gastrointestinal cancer patients? A phase 2 mixed-methods study. Palliat Med. 2018 Jan;32(1):46-58. doi: 10.1177/0269216317731571. Epub 2017 Sep 27. PMID 28952881